CLINICAL TRIAL: NCT06591962
Title: The Comparison of Biopsychosocial Characteristics of Individuals with Diabetes Mellitus and Without Diabetes Mellitus
Brief Title: The Comparison of Biopsychosocial Characteristics with and Without Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: Go 23/634
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; biopsychosocial model; BETY-BQ; validity and reliability; anxiety; depression
MeSH Terms: conditions — Diabetes Mellitus; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals diagnosed with diabetes mellitus: Individuals with diabetes mellitus admitted to the internal medicine outpatient clinic of a university hospital. A questionnaire will be applied for diabetes mellitus.
  Interventions: Other: Questionnaire application for diabetes mellitus
- Individuals without a diagnosis of diabetes mellitus: Individuals without diabetes mellitus admitted to the internal medicine outpatient clinic of a university hospital. A questionnaire will be applied for without diabetes mellitus.
  Interventions: Other: Questionnaire application for without diabetes mellitus

INTERVENTIONS:
Other: Questionnaire application for diabetes mellitus — Scales will be applied to individuals diagnosed with diabetes mellitus
  Groups: Individuals diagnosed with diabetes mellitus
Other: Questionnaire application for without diabetes mellitus — Scales will be applied to individuals diagnosed without diabetes mellitus
  Groups: Individuals without a diagnosis of diabetes mellitus

SUMMARY:
As it is a chronic disease, the lifelong disease duration and treatment process affect individuals with Type 2 Diabetes Mellitus (T2DM) biologically, psychologically, and socially by causing them to experience fatigue, increased stress, and life burden. Individuals with T2DM experience many psychosocial conditions leading to anxiety and depression as well as physical and functional effects. It has been reported that the fear of diabetic complications plays a vital role in depression, while individuals with diabetes with anxiety are more prone to depression. In addition, increased treatment cost burden has been reported among the psychological factors contributing to anxiety and depression in individuals with DM. One study reported that fatigue is commonly associated with increased anxiety, depression, and sleep problems in individuals with DM. A sedentary lifestyle in these individuals is noteworthy and has also been shown to be a contributing factor to depression.

In addition to improving diabetic complications due to the disease, reducing depressive states and improving the psychosocial status of individuals may positively affect diabetes and reduce the symptoms and complications of T2DM. It has also been reported that increasing the self-efficacy of individuals with diabetes may positively impact the treatment. Based on this information, it is clear that there is a need for physical and psychosocial evaluation of individuals with T2DM in disease management. Therefore, determination of the biopsychosocial effects of individuals with T2DM in improving disease-specific findings and quality of life of individuals with T2DM to reflect positively on disease management processes is necessary for holistic management in treating these individuals. However, studies in this field are insufficient. This study aimed to compare individuals with and without T2DM biopsychosocial characteristics.

The BETY-Biopsychosocial Questionnaire, which assesses the biopsychosocial status of individuals with rheumatism, has no validity in individuals with T2DM. Since the patient population and other scales to be used are common, it was considered to carry out the validity, reliability, and responsiveness study of this scale within the scope of this study.

ELIGIBILITY:
Individuals with Diabetes Mellitus

Inclusion Criteria:

* Being T2 DM
* To be between 18-65 years old

Exclusion Criteria:

* The patient has a diagnosis of autoimmune monogenic or drug-associated diabetes,
* Lack of consent of the participants,
* Frailty (Clinical Frailty Score; if greater than 3),
* Stroke, heart failure (NYHA stage 3 and above), unstable lung and cardiovascular diseases

Individuals without Diabetes Mellitus

Inclusion Criteria:

* Not having T2DM (other individuals followed up at Hacettepe University -
* Department of Internal Medicine)
* To be between 18-65 years old

Exclusion Criteria:

* The patient has a diagnosis of autoimmune monogenic or drug-associated diabetes,
* Lack of consent of the participants,
* Frailty (Clinical Frailty Score; if greater than 3),
* Stroke, heart failure (NYHA stage 3 and above), unstable lung and cardiovascular diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire | Three months
  The biopsychosocial status of the individual is assessed with questions about pain, functionality, mood, sociability, sexuality, and sleep status. Each question consists of 30 items scored between 0-120 as '0 (never), 1 (yes rarely), 2 (yes sometimes), 3 (yes often), 4 (yes always)'. A high score indicates poor biopsychosocial status.

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale (HADS) | Three months
  HADS consists of 14 items, 7 of which assess anxiety, and the other 7 determine depression. Each item is scored between 0-3, and the total is scored between 0-21. High scores indicate poor anxiety and depression levels.
Turkish version of the Multidimensional Diabetes Questionnaire | Three months
  The questionnaire consists of 3 sections, 7 sub-dimensions, and 41 items. Each section is evaluated separately; there is no total score for the scale.
  Section 1 focuses on the perception of diabetes and social support. It includes 16 items measured using a 7-point Likert-type scale.
  Section 2 evaluates the level of supportive and non-supportive behaviors of the diabetic spouse or caregiver towards self-care activities, using a 7-point Likert-type scale with 12 items.
  Section 3 assesses the perception of individual self-efficacy and outcome expectancy regarding managing the disease with 13 items measured on a Likert-type scale.
  High scores in perceived self-efficacy and outcome indicate a high level of expectation.
Summary of Diabetes Self-Care Activities | Three months
  The study participants were asked to report the frequency of their self-care activities, such as diet, exercise, blood glucose testing, foot care, and smoking, over the past seven days. They used a number line to indicate the number of days (between 0-7) for each activity, and smoking, they used a scale of 0 for nonsmokers and 1 for smokers, with an additional measure for the amount of cigarettes smoked. A higher score indicates a higher level of self-care activity.
Health Assessment Questionnaire (HAQ) | Three months
  The Health Assessment Questionnaire evaluates the functionality of the individual using eight parameters and 20 items. The parameters are classified as dressing, standing, eating, walking, hygiene, reaching, grasping, and other activities. Each item is scored as 0 (without any difficulty), 1 (with some difficulty), 2 (with a lot of difficulty), and 3 (unable to do at all). The total score is between 0-3, with a high score indicating low functionality.
General Health Questionnaire (Euro QoL-5D) | Three months
  The scale consists of 2 subsections. The first part, the EQ-5D-Index, consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to each dimension have three options; "no problem," "moderate problem," and "extreme problem." Index value results vary between "-0.59" and "1" points. "0" indicates death, and "1" indicates total health. Negative values indicate unconsciousness and bed dependency. The second part of the scale is the vertical visual analog scale (EQ-VAS), Which evaluates the subjective health perception of the individual between 0 and 100. Marked as the best health you can imagine and the worst health you can imagine.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will not be shared to protect the data of individuals